CLINICAL TRIAL: NCT01694628
Title: Psychosocial-Behavioral Therapy for Patients With Advanced COPD and Depression
Brief Title: Cognitive Behavioral Therapy for COPD
Acronym: CLIMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Lynn Foster Reinke, Clinical Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43252
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2016-10

CONDITIONS: COPD; Depression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLIMB (COPD Lifestyle, Mood, and Behavior) (Experimental): Counseling sessions for COPD and depression
  Interventions: Behavioral: CLIMB (COPD Lifestyle, Mood, and Behavior)
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: CLIMB (COPD Lifestyle, Mood, and Behavior) — Cognitive Behavioral Therapy delivered to patients via telephone aimed to improve mood and decrease depressive symptoms.
  Arms: CLIMB (COPD Lifestyle, Mood, and Behavior)

SUMMARY:
The purpose of this study in patients with advanced COPD and depression is twofold:

1. Determine the feasibility and acceptability of a 6-session e-counseling intervention
2. Determine the efficacy of the e-counseling intervention on depressive symptoms

We hypothesize that patients who participate in e-counseling will have improved depressive symptoms compared to patients receiving usual care at 8 weeks.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of the death in the US. Although COPD is mostly preventable, there is no cure. Thus, care of patients with COPD is primarily focused on symptom palliation with the goal of improving quality of life for both patients and their families. These goals are highly consistent with core principles of palliative care. Dyspnea is the most distressing symptom for patients. Even optimal disease-directed treatment provides only partial relief from dyspnea. Depression is consistently associated with worse dyspnea, but the mechanisms underlying this relationship are poorly understood. Since existing treatment for dyspnea has only limited success and there is evidence that treating depression alleviates pain, we propose that by improving mood, we may be more successful in alleviating dyspnea. Psychosocial-behavioral therapy (PBT) which is focused on increasing pleasant events and improving problem solving skills has been shown to have immediate and sustained effects on depressive symptoms in patients with dementia and post-stroke holds tremendous promise for efficacy in advanced COPD. Testing the use of novel technologies to provide efficacious interventions such as PBT to patients with advanced disease is critical for translational palliative care research

ELIGIBILITY:
Inclusion Criteria:

* COPD (FEV1/FVC < 70% & FEV1 <80%; current or past smoking >10pack-years)
* Depressed (PHQ-9 >=10)
* Ability to speak, read and write English
* Willingness to use computer or study-issued tablet device

Exclusion Criteria:

* Current non-nicotine substance abuse or dependence
* Psychotic disorder
* Active suicide ideation with intent and plan
* Alzheimer's/dementia
* Currently receiving any psychotherapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | 8 weeks
  Personal Health Questionnaire-9

SECONDARY OUTCOMES:
Dyspnea Intensity and Distress | 8 weeks
  Chronic Respiratory Questionnaire, Shortness of Breath Questionnaire, Dyspnea Management Questionnaire
Fatigue | 8 weeks
  Chronic Respiratory Questionnaire
Anxiety | 8 weeks
  Hospital Anxiety and Depression Scale
Physical Activity | 8 weeks
  Accelerometry (Stepwatch)
Quality of Life | 8 weeks
  Chronic Respiratory Questionnaire and Medical Outcomes Short Form-36

CONTACTS AND LOCATIONS:
Overall Officials: Lynn F Reinke, PhD, RN, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No